CLINICAL TRIAL: NCT02577887
Title: Advanced Bradycardia Device Feature Utilization and Clinical Outcomes II
Acronym: BRADYCARE II
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10073
Record Dates: First submitted 2015-10-06; First posted 2015-10-16 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Standard Bradycardia Pacing Indication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Patients implanted with a St. Jude Medical pacemakers

SUMMARY:
The purpose of this study is to characterize the utilization of diagnostics capabilities in St. Jude Medical pacemakers to manage patients with a standard bradycardia pacing indication.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, multi-center observational study designed to evaluate the utilization of diagnostic capabilities, indications, MRI scanning capabilities and clinical outcomes of patients implanted with SJM pacemakers.

The total duration of the study is expected to be approximately 30 months. The clinical study will be conducted in up to 160 centers across Europe, Middle East, Africa, (EMEA region) and Asia, Australia and New Zealand (Asia-Pac region). Approximately 2016 subjects will be enrolled in this study. Subjects will be followed for 1 year after pacemaker implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been implanted with an SJM Assurity MRI™, Endurity MRI™ or other SJM MRI compatible pacemakers in the EMEA region within 30 days or patients implanted with an Accent MRI™, Assurity MRI™, Endurity MRI™ or other SJM MRI compatible pacemakers in the Asia-Pac region within 30 days.
* Patient is geographically stable and willing to comply with the required follow-up schedule.
* Patient is not pregnant or planning to become pregnant during the course of the study.
* Patient is > 18 years of age

Exclusion Criteria:

* Patient's life expectancy is less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a standard bradycardia pacing indication and implanted with a St. Jude Medical pacemaker
Sampling Method: Non-Probability Sample
Enrollment: 2101 (Actual)
Dates: Start 2015-07; Primary Completion 2017-11-25 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, Study Director — Abbott Medical Devices
Locations (4):
- 114 Avenue d'Arès, Bordeaux, France
- Kliniken der Friedrich-Alexander-Universität, Erlangen, Germany
- Via Palermo 636, Catania, Italy
- 2-15 Yamadaoka, Suita, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Consented Patients: Patients implanted with Accent MRI, Assurity MRI, Endurity MRI or other newer SJM pacemakers, with a standard indication for implant.
Period: Overall Study
Arm/Group | All Consented Patients
Started | 2101
6 Month Follow-up | 1938
Completed (The last follow-up was at 12 months post implant.) | 1803
Not Completed | 298
Not completed — Death | 93
Not completed — Protocol Violation | 125
Not completed — Withdrawal by Subject | 80

BASELINE CHARACTERISTICS:
Population: All consent patients.
Arm/Group | All Consented Patients
Number analyzed (Participants) | 2101
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 896
  Male | 1205
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 234
  Italy | 178
  France | 241
  Germany | 236
  Austria | 96
  Belgium | 64
  China | 48
  Estonia | 183
  Finland | 92
  Hong Kong | 10
  India | 56
  Lithuania | 46
  Netherlands | 131
  Portugal | 102
  South Korea | 155
  Spain | 157
  United Kingdom | 72
Primary Indication [Count of Participants; unit: Participants]
  Sinus Node Dysfunction | 868
  AV Node Block | 1026
  Syncope | 189
  Prevention/Termination of Tachyarrhythmias by Paci | 16
  Pacemaker replacement | 2
Cardiovascular History [Count of Participants; unit: Participants]
  Angina | 62
  Cardiomyopathy | 438
  Coronary Artery Disease | 452
  Heart Failure | 4
  Hypertension | 1371
  Myocardial infarction | 182
Medication [Count of Participants; unit: Participants]
  ACE Inhibitors/ ARBs | 1124
  Aldosterone Inhibitors | 85
  Anti-Coagulants | 679
  Antiarrhythmics- Class I | 82
  Antiarrhythmics- Class III | 98
  Antiplatelet | 665
  Beta Blockers | 711
  Calcium Channel Blockers | 612
  Cardiac Glycosides | 46
  Diuretics | 730
  Nitrates | 109
  Other Cardiac | 96
  Positive Inotropics | 3
  Statins | 154
Blood Pressure (mm Hg) [Mean (Standard Deviation); unit: mm Hg]
  Diastolic Blood Pressure | 74.8 (12.2)
  Systolic Blood Pressure | 138.3 (21.9)
Ejection Fraction (%) [Mean (Standard Deviation); unit: % of blood leaving heart at contraction] | 59.6 (9.4)
Heart Rate (bpm) [Mean (Standard Deviation); unit: bpm] | 64.2 (16.4)
Other Medical History [Count of Participants; unit: Participants]
  Diabetes | 509
  Heaptic/Renal disease | 253
  Peripheral vascular disease | 90
  Pulmonary disease | 89
  Smoking | 634
  Stroke | 216
Cardiovascular Interventions [Count of Participants; unit: Participants]
  Ablation | 3
  Coronary Artery Bypass Grafting (CABG) | 113
  Perc Coronary Intervention (PCI )/ Atherectomy | 251

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complications in the General Pacemaker Population
Description: The rate of device related adverse events that require a medical intervention and/or hospitalization for treatment.
Time Frame: 1 year
Population: All subjects.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | All Consented Patients
Number analyzed (Participants) | 2101
percentage of subjects | 3.33 [2.6 to 4.2]

2. Secondary Outcome: Number of Subjects Programmed With Advanced Pacemaker Features
Description: Advanced pacemaker features include Autocapture, Auto sensitivity control (ASC), Ventricular Intrinsic Preference (VIP®), Patient Notifier, RF telemetry, and newer advanced features.
Time Frame: 1 year
Population: All study participants that completed that 12-month visit and had the feature enabled for the duration of the study. Subjects that had a change in the status of the feature (e.g. ON to OFF) are not included in the count shown here.
Measure: Count of Participants; unit: Participants
Arm/Group | All Consented Patients
Number analyzed (Participants) | 1803
Participants
  Ventricular Intrinsic Preference | 732
  AF Suppression | 10
  Trigger Alert: High RV Rate: number analyzed (Participants) | 1798
  Trigger Alert: High RV Rate | 1738
  Trigger Alert: High V Rate during AT/AF: number analyzed (Participants) | 1798
  Trigger Alert: High V Rate during AT/AF | 1439
  Trigger Alert: AT/AF: number analyzed (Participants) | 1798
  Trigger Alert: AT/AF | 1432
  Trigger Alert: Exceeded AT/AF Burden: number analyzed (Participants) | 1798
  Trigger Alert: Exceeded AT/AF Burden | 1433
  Trigger Alert: % V Pace: number analyzed (Participants) | 1798
  Trigger Alert: % V Pace | 1280
  Trigger Alert: Atrial Impedance Out of Range: number analyzed (Participants) | 1798
  Trigger Alert: Atrial Impedance Out of Range | 34
  Trigger Alert: Ventricular Impedance Out of Range: number analyzed (Participants) | 1798
  Trigger Alert: Ventricular Impedance Out of Range | 37
  Remote Monitoring | 198
  Atrial Capture Confirm | 245
  Right Ventricular Auto Capture | 678
  Atrial Pace during PMT | 1412

3. Secondary Outcome: Number of Pacemaker Patients With Atrial Tachycardia/Fibrillation (AT/AF), Ventricular Tachycardia/Fibrillation (VT/VF), Pacemaker-mediated Tachycardia (PMT) and Automatic Mode Switching (AMS) Episodes
Description: At each follow-up, devices were interrogated and device session records were uploaded. Episodes of AT/AF, VT/VF, PMT and AMS were measured by the pacemakers diagnostics features.
Time Frame: 1 year
Population: All patients that completed the 12-month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | All Consented Patients
Number analyzed (Participants) | 1803
Participants
  Number of subjects with PMT | 563
  Number of subjects with AT/AF | 427
  Number of subjects with VT/VF | 861

4. Secondary Outcome: Number of MRI Scans by Country
Description: The total number of scans performed by country
Time Frame: 1 year
Population: All study participants
Measure: Number; unit: scans
Arm/Group | All Consented Patients
Number analyzed (Participants) | 2101
scans
  Estonia | 34
  Italy | 14
  Germany | 13
  Japan | 13
  France | 10
  Belgium | 7
  Austria | 6
  Netherland | 5
  Spain | 4
  South Korea | 4
  Finland | 2
  UK | 2
  Portugal | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | All Consented Patients
All-Cause Mortality (participants affected / at risk) | 94/2101
Serious Adverse Events (participants affected / at risk) | 70/2101
Other Adverse Events (participants affected / at risk) | 19/2101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Consented Patients (N=2101)
Loss of Normal Desired Pacing and/or Sensing due to Lead Displacement (Product Issues) | 25 (26)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Unknown Death (General disorders) | 6 (6)
Cardiac Perforation (Injury, poisoning and procedural complications) | 4 (4)
Hematoma (Vascular disorders) | 4 (4)
Lead Malfunction (Product Issues) | 3 (3) — Fracture or damage to insulation
Arrhythmia (Cardiac disorders) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Cardiac Tamponade (Cardiac disorders) | 2 (2)
Endocarditis (Cardiac disorders) | 2 (2)
Pacemaker Mediated Tachycardia (Product Issues) | 2 (2)
TIA (Nervous system disorders) | 2 (2)
Device Migration (Injury, poisoning and procedural complications) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Inflammatory Allergic Reaction (Immune system disorders) | 1 (1)
Lead Misplacement (Injury, poisoning and procedural complications) | 1 (1)
Loss of Normal Device Function due to Battery Failure or Component Malfunction (Product Issues) | 1 (1)
Pericarditis associated with Dressler's Syndrome (Cardiac disorders) | 1 (1)
Pocket Erosion (Injury, poisoning and procedural complications) | 1 (1)
Reduction of LVEF due to RV Pacing (Investigations) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Threshold Elevation (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Consented Patients (N=2101)
Hematoma (Vascular disorders) | 5 (5)
Arrhythmia (Cardiac disorders) | 3 (3)
Lead Noise (Product Issues) | 3 (3)
Threshold Elevation (Product Issues) | 3 (3)
Extracardiac Stimulation (Product Issues) | 2 (2)
Pacemaker Mediated Tachycardia (Product Issues) | 2 (2)
Pain at IPG Site (General disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT02577887/Prot_SAP_000.pdf